CLINICAL TRIAL: NCT05927272
Title: Deciphering the Vitiligo Transcriptomic Signature Between Repigmented and Non Repigmented Lesions
Acronym: STRAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2021/54
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: monocentric, open-label study, and translational research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with active non-segmental vitiligo (Experimental)
  Interventions: Procedure: SKIN SAMPLES; Procedure: BLOOD SAMPLES; Device: narrowband UVB; Drug: Systemic Steroids

INTERVENTIONS:
Procedure: SKIN SAMPLES — At baseline: one 4 mm Ø skin biopsies: on forearms (excluding skin folds): fresh At month 3 and month 6: Two 4 mm Ø skin biopsies will be performed on the same lesion selected at baseline (one on a repigmented area, one on a non-responded area): fresh
  Fresh Skin biopsies will be analyzed the same day using Single-cell RNA sequencing (scRNAseq).
Procedure: BLOOD SAMPLES — Blood samples will be taken (30 mL) at week 0, week 12, week 24 for the measurement of pro-inflammatory cytokines and chemokines ligands in blood sera.
Device: narrowband UVB — narrowband UVB (Nb-UVB) 2 times a week
Drug: Systemic Steroids — Oral minipuls of systemic steroids (Medrol 16mg twice a week) for 24 weeks

SUMMARY:
The purpose of this study is to perform an in-depth analysis of the molecular pathways involved in lesions responding to current treatment and lesions not responding to current treatment

DETAILED DESCRIPTION:
Treatment strategy: combination of oral mini-pulse of methylprednisolone 16mg twice a week + phototherapy Ultraviolet B (UVB) TL01, 2 times a week.

One skin biopsy will be performed at baseline and two skin biopsies at month 3 and month 6 on the same area forearms (excluding skin folds) Blood samples will be taken (30 mL) at week 0, week 12, week 24 for the measurement of pro-inflammatory cytokines and chemokines ligands in blood sera.

Principal Objective:

The aim of this study is to perform an in-depth analysis of vitiligo skin and blood samples taken during the course of a standard therapy to identify pathways involved in the repigmentation.

Secondary Objectives:

* Evolution of Vitiligo Disease in relation of patient profile
* Evolution of the activity of vitiligo in relation of patient profile The statistical and bioinformatics analyzes will be carried out on the data resulting from research with correlation to clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Subject: male or female aged ≥ 18 years and ≤ 65 years
* Diagnosis of non-segmental (symmetrical) vitiligo with a body surface area involved >5% excluding hands and feet, with lesions located on arms
* Active non-segmental vitiligo is defined by:

  * Non-segmental vitiligo with new patches or extension of old lesions during the last 6 months AND
  * Presence of hypochromic aspect under Wood's lamp examination and/or perifollicular hypopigmentation under Wood's lamp examination.
* Able to read, understand, and give documented informed consent
* Registered in the French Social Security
* Patients that could receive the combination of oral steroids and phototherapy according the recommendation
* Signed informed consent form

Exclusion Criteria:

* Segmental or mixed vitiligo
* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.
* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-10-09 (Estimated); Study Completion 2025-10-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the evolution of skin biological pathways, assessed by single cell RNAseq in the peri-lesional and lesional skin of a target lesion | Month 6
  Identify pathways involved in the repigmentation using transcriptomic analyses with Single-cell RNA sequencing (scRNA-seq), comparing molecular/cellular background between vitiligo skin lesions responding to current treatment and lesions not responding to current treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Julien SENESCHAL, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux - St André Hospital, Bordeaux, France